CLINICAL TRIAL: NCT02761434
Title: The Effect of Osmotically Stimulated Vasopressin on Glucose Regulation
Brief Title: The Effect of Vasopressin on Glucose Regulation
Acronym: HYPERGlu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Stavros Kavouras, Associate Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-12-360
Record Dates: First submitted 2016-04-26; First posted 2016-05-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Insulin Resistance
Keywords: copeptin; vasopressin; dehydration; insulin resistance; Diabetes; Glucose regulation
MeSH Terms: conditions — Insulin Resistance; Diabetes Insipidus; Dehydration; Diabetes Mellitus | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dehydration (Active Comparator): Infusion of 3% sodium chloride for osmotic stimulation of vasopressin
  Interventions: Other: Hypertonic Saline (3% NaCl)
- Euhydration (Placebo Comparator): Infusion of 0.9% sodium chloride that will induce similar expansion of plasma volume without any significant change in osmolality and vasopressin
  Interventions: Other: Isotonic Saline (0.9% NaCl)

INTERVENTIONS:
Other: Hypertonic Saline (3% NaCl) — 0.1 ml of 3% NaCl per kg of body weight per minute
  Arms: Dehydration
Other: Isotonic Saline (0.9% NaCl) — 0.1 ml of 0.9% NaCl per kg of body weight per minute
  Arms: Euhydration

SUMMARY:
Data from experimental animals and human epidemiological studies have suggested that hypohydration and/or low water intake is linked to poor glucose regulation and diabetes. The aim of this study is to investigate the effects of cellular dehydration on glucose in healthy non-diabetic individuals. METHODS: 60 males and females (30-55 y) will will undergo two experimental trials (ISO and HYP), consisting of a 2-h intravenous infusion of isotonic or hypertonic saline on two separate occasions, followed by a 4-h oral glucose tolerance test. Blood samples were taken from an antecubital vein in 30-min intervals starting at baseline for assessment of fluid and glucose regulating factors. Thirst will be assessed via visual analog following each blood sample. Energy substrate oxidation will be calculated via indirect calorimetry every 60 min.

DETAILED DESCRIPTION:
Introduction The neurohypophysial hormone arginine vasopressin (AVP), also known as antidiuretic hormone, was one of the first hormone identified for its vasopressin properties in 1895 by Oliver and Schäfer. They showed that extract of pituitary gland increased blood pressure in anesthetized dogs. AVP is mainly synthesized in the paraventricular and supraoptic nucleus of the hypothalamus. The hormone is transferred to the neural lobe of the posterior pituitary where it is released to the circulation. Target organs perceive the hormonal stimuli by three different receptors: V1a, V1b and V2. The receptor V1a is mainly expressed in the vascular wall and is responsible for vasoconstriction. The receptor V1b is mainly found in the anterior pituitary, mediating the secretion of the adrenal corticotropin hormone, while the V2 receptor is mainly expressed in nephron tubules triggering water reabsorption. Since the discovery of AVP, both the vasopressin and antidiuretic properties have been very well studied and documented.

Other than the AVP effects on blood pressure and water homeostasis, the hormone is implicated in a variety of other functions including pain, bone and lipid metabolism, hypertension, social behavior, aging, cognitive function, cellular proliferation, inflammation, infections, homeostasis, hypothalamic-pituitary-adrenal axis, and diabetes. All these effects could provide useful insight into many diseases. Therefore, the focus of this application is on the effects of AVP on glucose regulation in healthy humans.

AVP is known to enhance hepatic glycogenolysis by activation of V1a receptors and by increasing the release of glucagon, resulting in increased glucose levels in experimental animals. Even when glucagon receptors in the liver are blocked, AVP still increases blood glucose. The V1b receptors have been identified in both alpha and beta cells of the islets of Langerhans. Thus, AVP stimulates insulin secretion counteracting the increase in blood glucose. In an experiment with AVP V1a and V1b receptor knockout mice, alterations in glucose and fat metabolism were observed, suggesting that AVP might play a role in glucose regulation and metabolic disorders. Studies in humans with a genetic variation of AVP V1a receptor showed increased prevalence of diabetes in overweight or subjects with high fat diet. Recently, a study in rats prone to metabolic dysfunction, examined the effect of long-term influence of vasopressin on glucose homeostasis. It reported that high vasopressin enhanced hyperinsulemia and glucose intolerance in obese rats, while treatment with vasopressin receptor V1a antagonist reduced glucose intolerance.

In a French epidemiological study, a cohort of 3,615 males and females with normal fasting blood glucose was followed for 9 years. It indicated that water intake was inversely and independently associated with the risk of developing hyperglycemia. The authors hypothesized that their results were due to hypohydration related increase in plasma vasopressin. More recently, a Swedish cohort of 2,064 subjects from the malmo diet and cancer study was analyzed after 15.8 y with an oral glucose tolerance test. They found that copeptin (a reliable and clinical surrogate marker of AVP) independently predicted diabetes mellitus and abdominal adiposity.

Interestingly, hypohydration and low water drinking is linked to chronic elevated AVP. In a recent study with free-living adults, low habitual water intake led to significantly elevated AVP compared to adults with high water intake.

Experimental Design Sixty subjects between the age of 30 to 55 with absence of insulin resistance will be recruited in the study. Thirty of the adults will be with normal body mass index (BMI; 15 males and 15 females, 18.5 kg∙m-2 < BMI ≤25 kg∙m-2) and thirty overweight or obese adults (15 males and 15 females, 28 kg∙m-2 ≤ BMI ≤35 kg∙m-2) will be recruited to participate in the study. Sample size estimation showed that 60 subject will provide power of 0.8 with alpha level set at 0.05. The effect of vasopressin on glucose metabolism will be studied via osmotic stimulation of vasopressin (AVP) utilizing hypertonic saline infusion followed by an oral glucose tolerance test. Each subject will perform two identical experiments, differing only in the sodium chloride (NaCl) content of the infusion (isotonic vs. hypertonic saline). All female subjects will perform both trials during their early follicular phase, approximately 2-6 days post menses onset to ensure low endogenous levels of estrogen and progesterone. After resting in a seated position for 30 min, subjects will be infused intravenously either 3% NaCl (Hypertonic saline, hence HYPER) or 0.9 % NaCl (Isotonic saline, hence ISO) over a 120 min period at an infusion rate 0.1 ml/min/kg of body weight in a single-blind fashion and in counterbalanced order. This hypertonic saline infusion increases plasma osmolality from 285 to at least 300 mmol/kg. From a separate venous catheter, blood samples will be taken every 30 min. Following infusion, subjects will rest for an equilibration period of 30 min before they start a 4-h oral glucose tolerance test.

Subject preparation for oral glucose tolerance test (OGTT): Subjects should eat a normal diet for 3 days prior to the test, and undertake normal physical activity. Dinner will be standardized the day before and no alcohol will be allowed. Subjects will be instructed to fast at least 10 h prior to the test.

Procedure for OGTT: The OGTT test will consist of a 75 g of glucose ingestion followed by blood sampling period, with samples collected every 30 min for 240 min. Urine samples will be collected at the end of the infusion and at the end of the OGTT. Blood pressure will be recorded via an automated sphygmomanometer following each blood sample. Oxygen uptake and respiratory exchange rate will be assessed hourly via indirect calorimetry, for a total of seven times per trial. During blood sampling, thirst perception and mouth dryness will be also assessed via visual analog scales.

Samples Analysis A total of fourteen blood samples will be collected in each experimental trial and analyzed for: hematocrit (Hct), hemoglobin (Hb), osmolality (Osm), sodium (Na) and potassium (K), total plasma protein, glucose, insulin, c-peptide, glucagon, copeptin, plasma renin activity, corticotropin releasing hormone (CRF), cortisol, triglycerides and free fatty acids (FFA).

Urine samples will be analyzed for osmolality and urine specific gravity fresh. Backup samples of serum, plasma, and urine will be stored, frozen at -80°C, in the event additional analysis are needed, or as replacements for broken vials.

Data Handling & Analysis To ensure quality and integrity of the data collected case report forms will be utilized. The case report forms (CRF) will be designed to record data collected in a way that will meet the highest standards. CRF will be developed, tested and approved prior to any subject enrolment. The scientist involved in the data collection of the study will be trained on the use of CRF prior to beginning of data collection. A paper and digital library for all CRFs will be established and maintained during the experiment and at least for 2 more years after the publication of the manuscripts. The data base manager and the principal investigator will be the only person that will have access to identifiable subject information. All the rest of the documents will be coded to ensure subject anonymity. Data and Safety Monitoring Plan includes: Overall framework for data and safety monitoring, responsible party for monitoring, and procedures for reporting adverse events/unanticipated problems. Following data collection, data entry will take place by two authorized scientists. Data from Quest diagnostics are available in PDF format and data entry will be also performed and verified by two scientists. Data integration and database cleaning will be performed in statistical software via analysis and visualization.

The primary response variable glucose metabolism will be captured by 4 variables (glucose, insulin, C-Peptide and glucagon) all measured on a ratio scale, and on 14 occasions.

Secondary Outcomes will be: Hb, Hct, Total Proteins, Osmolality, Na, K, Copeptin, adrenal corticosteropin releasing hormone (ACTH), CRH, Angiotensin II, plasma renin activity (PRA), Aldosterone, Triglycerides, FFA.

Additional repeated continuous outcomes will be: (1) Blood pressure which will be measured on 14 occasions; (2) Oxygen uptake and respiratory exchange rate which will be assessed on 7 separate occasions; and (3) thirst perception and mouth dryness which will be measured on 14 occasions.

Covariates Measurements Treatment groups (isotonic vs. hypertonic saline) will be the primary comparison of interest. Other covariates will include sex (Females vs. males) and weight status (normal weight vs. overweight/obese), age (30-55) and time (1-14).

To examine if the mean response profiles are similar in the groups, i.e. whether patterns of change over time in the mean response vary by group, the present study will further explore group by time interaction effects: (e.g. treatment by time interaction; weight by time interaction; sex by time interaction).

Data Analysis Plan

* For this quasi-experimental with repeated measure-design, the researchers will conduct a longitudinal analysis to describe changes in the mean response over time, and how these changes are related to the covariates of interest.
* The normality of these continuous variables will be assessed by conducting the Shapiro-Wilk test of normality.
* For all continuous outcomes, summary statistics (mean and standard deviations) will be conducted at each time and by sequence. Moreover, correlations between glucose metabolism measures will be performed.
* Percentages will be calculated for covariates that are measured on a nominal scale, and mean and ± standard deviations presented for those measured on a continuous scale.
* The distributions of insulin sensitivity indexes and areas under the curve will be will be assessed.

Statistical Modeling To study how changes in the mean response relate to covariates over time, Generalized Linear Mixed Effects Modeling -with random intercepts and slopes- will be employed using the Restricted Maximum Likelihood Estimation. It is assumed that each group's mean response will change linearly over time. However, if the mean response over time is not linear, higher-order polynomial trends will be explored.

The researcher will fit the appropriate covariance pattern model to account for the correlations among the repeated measures so that appropriate inferences are made.

Statistical significance will be determined at an alpha of 0.05. All statistical analyses would be carried out with the following statical software STATA©, JMP© or SAS©.

Anticipated Findings and Conclusions During the hypertonic saline infusion trial water balance will be artificially manipulated (hypertonic hypervolemia). The increase in plasma osmolality will stimulate vasopressin secretion. It is anticipated that AVP stimulation will elevate insulin to a greater degree than glucose resulting in higher insulin resistance. It is also expected that great urine osmolality as a response to elevated vasopressin levels and lower urinary output.

Significance of the Project Diabetes along with obesity is one of the leading non-communicable diseases in the developed and developing countries. More than 29 million Americans are diabetic and another 86 million are in a pre-diabetic state. The cost of diabetes in 2012 was $245 billion and it is growing. Hypohydration on the other side, is a quite common phenomenon linked to many health issues like urinary tract infections, kidney stones, cardiovascular diseases, mood state and cognitive performance. One of the potential mechanisms behind the effects of hypohydration is the elevated level of AVP. Recent epidemiological data and experiments in animals indicate that hypohydration and high vasopressin are linked to both diabetes and glucose dysregulation. However, no experimental data from a controlled trial in humans exist. The purpose of the proposed study is to perform a controlled trial on healthy humans to examine the effect of elevated vasopressin on glucose regulation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of age 30-50 y old
* Signed Informed Consent prior to the initiation of any trial procedure
* Sedentary lifestyle

Exclusion Criteria:

* Body Mass Index (BMI) greater than 35 kg/m2, below 18.5 kg/m2, and between 25 and 28 kg/m2
* Surgical operation on digestive tract, except possible appendectomy
* Regular smoker within the past 6 months
* Diagnosed diabetes (Type I or Type II)
* Previous diagnosis of cardiovascular disease including hypertension
* Inability to participate in the entire study
* Drastic change in weight in the last month (more than 3 kg)
* Serotonin re-uptake inhibitors (i.e. Prozac)
* Impaired kidney or liver function
* Insulin therapy
* injectable contraceptives
* Currently taking medications that impair water balance
* Commuting by bike the day of the experiment
* Pregnancy

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Glucose area under the curve during the 4 h following ingestion of 75 g glucose | Within 4 hours of the hypertonic saline infusion
  the area under the glucose curve (AUC) in mg/dL x min
Insulin area under the curve during the 4 h post ingestion following ingestion of 75 g glucose | Within 4 hours of the hypertonic saline infusion
  the area under the insulin curve (AUC) in microU/mL x min
Insulin sensitivity by matsuda & quicki Index | Within 4 hours of the hypertonic saline infusion

SECONDARY OUTCOMES:
Thirst, mouth dryness | during the experiment every 30 min for the 6 ½ hours of the experiment
  the response of thirst and mouth dryness will be scored in mm via a visual analog scale of 125mm length.
Resting metabolic rate | every 60 min of the experiment for the 6 ½ hours of the experiment
  Energy expenditure calculated via indirect calorimetry in kcal/min
Energy substrate oxidation | every 60 min of the experiment for the 6 ½ hours of the experiment
  g of carbohydrates and fat oxidized based on the amount of oxygen consumed and carbon dioxide produced assessed by indirect calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

REFERENCES:
- [Derived] Jansen LT, Suh H, Adams JD, Sprong CA, Seal AD, Scott DM, Butts CL, Melander O, Kirkland TW, Vanhaecke T, Dolci A, Lemetais G, Perrier ET, Kavouras SA. Osmotic stimulation of vasopressin acutely impairs glucose regulation: a counterbalanced, crossover trial. Am J Clin Nutr. 2019 Dec 1;110(6):1344-1352. doi: 10.1093/ajcn/nqz236. PMID 31562496